CLINICAL TRIAL: NCT03057392
Title: The Effect of Head Out Water Immersion During Dialysis on Clinical Parameters, Hemodynamic Parameters, and Hormonal Parameters in 10 Hemodialysis Patients
Brief Title: Head Out Water Immersion for Hemodynamic Stability During Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 73/12
Record Dates: First submitted 2014-06-11; First posted 2017-02-20 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Intradialytic Hypotension; Immersion
Keywords: immersion; ultrafiltration; dialysis
MeSH Terms: interventions — Immersion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- immersion and them sham procedure (Experimental): hemodialysis patients will do a 3 hours dialysis session while sitting in a bath and then have a "dry session" outside the bath
  Interventions: Other: immersion
- sham session and then immersion (Sham Comparator): dialysis patients will have a 3 hour dialysis session (dry session) and then immersion
  Interventions: Other: sham session

INTERVENTIONS:
Other: immersion — participants will sit in a 34-35C while receive dialysis
  Arms: immersion and them sham procedure
Other: sham session — dialysis while sitting in the dialysis chair
  Arms: sham session and then immersion

SUMMARY:
Immersion to the neck before and during hemodialysis session may increase intravascular volume, potentiate the ability to ultrafiltrate excess water, with less symptoms of shock, muscle crumps etc.

The aim of the present study is to compare blood volume, hemodynamic and endocrine parameters of chronic ESRD patients undergoing forth dialysis session in water immersion vs. control regular session.

DETAILED DESCRIPTION:
10 chronic hemodialysis patients, treated in the hemodialysis unit of Asaf-Harofeh Medical Center will be enrolled in the study.

Hemoglobin and albumin will be detected at baseline, and a recent (less than one year) echo will be used for the detection of ejection fraction.

The study will be a cross over study. Each set of studies will consist of two dialysis sessions, an immersion session, and a dry, non-immersion session. The study sessions will be short, 3 hours sessions with 250-350 ml/min blood flow (depends on the patients access) dialysate flow was 500 ml/min and dialysate sodium was 137meq/l. The temperature of the dialysate will be adjusted to 37°C and its composition as follows: Na+ = 137 mEq/L, K+ = 2.0 mEq/L, Ca2+ = 3.0 mEq/L, Mg2+ = 1.0 mEq/L, HCO3-= 30 mEq/L, glucose =100 mg/dL, CH3COO-= 8 mEq/L. The sodium concentration will be constant during treatment.

Ultrafiltration will be determined as the mean of UF during the ten previous sessions±10% according to the patients weight on admission. The immersed and dry session will be done in the midweek sessions, in random order, at least one week apart from each other.

Head-Out Water Immersion

A bath will be used for immersion. The bath will be filled with purified water before each of the session, and will be heated to 34-35°C. Patients will enter the bath and sat upright for few minutes and then connected to dialysis. The water will circulate through a thermostats and heating device in order to maintain a constant temperature.

Patients with arterio-venous fistula or graft in their arm will be immersed in water up to their axilla, with their arm lining on a floating pad. For patients with perm-cath immersion will only be done up to 5 cm below the catheter insertion.

Study procedure

Subjects will enter the bath and sit for few minutes, after which blood samples will be drown for baseline measurement. During the session blood pressure and heart rate will be measured every 15 minutes by conventional sphygmomanometry. and blood volume will be estimated by using blood volume monitor (Crit-Line).

Blood samples will be drown at baseline and after one hour, and before caseation of the session for plasma renin activity, aldosterone, atrial natriuretic peptide. Baseline and end of session urea will also measured for URR.

ELIGIBILITY:
Inclusion Criteria:

* chronic hemodialysis patients

Exclusion Criteria:

* anemia (HB<10) active infectious disease cognitive impairment dialysis access installed in the leg inability to cooperate with the study procedure Clinically evident overhydrated patients(edema, pulmonary congestion, pulmonary effusion)

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
symptomatic hypotension during dialysis | 3 hours
  a decrease of systolic BP of 22mmHG or more or decrease of diastolic BP of 10 mmHg or more accompanied with symptoms of muscle crumps, presyncope or syncope

SECONDARY OUTCOMES:
blood pressure changes compared to baseline | 3 hours every 15 min
  analysis by electronic sphygmomanometer every 15 minutes during the session
Atrial natriuretic peptide change compared to baseline | 0, 1, 3 hours
  blood will be drown from arterial line at baseline, after one hour and after 3 hours before dialysis termination.

CONTACTS AND LOCATIONS:
Locations (1):
- Dialysis Clinic in Asaf Harofhe Medical Center, Ẕerifin, Israel